CLINICAL TRIAL: NCT01994447
Title: "Traditional Research Nurses Versus an Innovative Undergraduate Research Assistant Program: Parental Understanding of Informed Consent " (the TRAIN Study)
Brief Title: The Train Study: Parental Understanding of Informed Consent
Acronym: TRAIN
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Change in study consent process at study site so that study had to be terminated
Sponsor: University of Calgary (Other)
Responsible Party: Principal Investigator, Antonia Stang, Assistant Professor, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: ACHF-001
Record Dates: First submitted 2013-11-19; First posted 2013-11-25 (Estimated); Last update posted 2016-10-26 (Estimated); Status verified 2016-10

CONDITIONS: Parental Comprehension of Informed Consent
Keywords: Informed Consent; Instructional Films and Video; Consent Comprehension; Multimedia Consent; Parent

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Traditional Nurse Enrollment (No Intervention): Research nurses will obtain verbal consent from patient/caregiver.
- Student Enrollment (Experimental): Trained research students will use digital video discs (DVD's) of primary investigators explaining study information to obtain informed consent
  Interventions: Other: Student Enrollment

INTERVENTIONS:
Other: Student Enrollment — The standard informed consent process is for research nurses to provide verbal explanations of studies. In the intervention arm trained research students will use DVD's made by the studies principal investigator to explain study information in the informed consent process.
  Arms: Student Enrollment

SUMMARY:
Project Summary: One of the challenges facing pediatric researchers is the need to balance decreasing funding with the time and human resource costs associated with enrolling children. In order to address this, the Emergency Department (ED) research team developed an innovative model for subject enrollment and consent using highly trained and supervised undergraduate students. From a human resources perspective, utilizing students is more cost effective than the traditional research nurse model. However, a concern with this method is the adequacy of parental understanding of study information for informed consent. The aim of this project is to determine if the use of students is at least as good as the more costly "gold standard" of experienced research nurses. The validation of this innovative student model will enable child health investigators to better meet parent's needs and increase the efficiency of pediatric research.

The primary objective of this study is to measure parental comprehension of informed consent information using an innovative undergraduate research assistant program compared to consent using the traditional research nurse model. We hypothesize that parental comprehension of the informed consent information process when approached by undergraduate students will be comparable (or not worse) than when consent is obtained by a research nurse.

ELIGIBILITY:
Inclusion Criteria:

* Parent's child must be eligible for an interventional study in the Alberta Children's Hospital Emergency Department
* Parent or accompanying adult must be the legal guardian
* One independent trained research student and one research nurse must be available for randomization
* Parent must be exposed to entire informed consent process

Exclusion Criteria:

* Previous participant in the TRAIN study
* Parental language barrier

Max Age: 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 12 (Actual)
Dates: Start 2013-11; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Parental understanding of informed consent process using a standardized measurement tool, the Deaconess Informed Consent Comprehension Test (DICCT) | 1 day ED visit
  The DICCT is a validated and reliable tool that was developed to assess comprehension of informed consent information among adult study subjects and adapted to measure parental understanding of consent. Parental understanding of the consent process will be measured using a modified Deaconess Informed Consent Comprehension Test (mDICCT), which has previously been used in a pediatric setting. The score on the DICCT will be presented as a mean or median (depending on distribution) with 95% Confidence Intervals (CI's). The appropriate parametric (t-test) or non-parametric test will be used to compare the score on the DICCT between the intervention (student enrollment) and the control group (traditional nurse enrollment).

SECONDARY OUTCOMES:
Duration of consent process | 1 day ED visit
  Duration of consent process from initial approach to time consent form is obtained or consent refused will be reported for all enrolled patients (median, IQR) as well as for patients in the intervention (student enrollment) and control group (traditional nurse enrollment).
Length of stay of the patient in the department | 1 day ED visit
  Length of stay in the ED for all patients enrolled in the study, for patients in the intervention group (student enrollment) and in the control group (traditional nurse enrollment), presented as medians with IQR.

OTHER OUTCOMES:
consent rate | 1 day ED visit
  Proportion of patients/caregivers who consent in the intervention (student enrollment group) and in the control (traditional nurse enrollment) group reported as a proportion with 95% CI's.

CONTACTS AND LOCATIONS:
Overall Officials: Antonia S Stang, MD, Principal Investigator — Department of Pediatrics, University of Calgary
Locations (1):
- University of Calgary, Alberta Children's Hospital Emergency Department, Calgary, Alberta, Canada

REFERENCES:
- [Background] Davis DP, Poste JC, Kelly D. The UCSD Research Associate Program: a recipe for successfully integrating undergraduates with emergency medicine research. J Emerg Med. 2005 Jan;28(1):89-93. doi: 10.1016/j.jemermed.2004.07.012. PMID 15657015
- [Background] Hollander JE, Singer AJ. An innovative strategy for conducting clinical research: the academic associate program. Acad Emerg Med. 2002 Feb;9(2):134-7. doi: 10.1111/j.1553-2712.2002.tb00230.x. PMID 11825839
- [Background] Miller CK, O'Donnell DC, Searight HR, Barbarash RA. The Deaconess Informed Consent Comprehension Test: an assessment tool for clinical research subjects. Pharmacotherapy. 1996 Sep-Oct;16(5):872-8. PMID 8888082
- [Background] Tait AR, Voepel-Lewis T, Malviya S. Do they understand? (part I): parental consent for children participating in clinical anesthesia and surgery research. Anesthesiology. 2003 Mar;98(3):603-8. doi: 10.1097/00000542-200303000-00005. PMID 12606901
- [Background] Segal S, Lloyd T, Houts PS, Stillman PL, Jungas RL, Greer RB 3rd. The association between students' research involvement in medical school and their postgraduate medical activities. Acad Med. 1990 Aug;65(8):530-3. doi: 10.1097/00001888-199008000-00010. PMID 2383337
- [Background] Ryan RE, Prictor MJ, McLaughlin KJ, Hill SJ. Audio-visual presentation of information for informed consent for participation in clinical trials. Cochrane Database Syst Rev. 2008 Jan 23;(1):CD003717. doi: 10.1002/14651858.CD003717.pub2. PMID 18254029
- [Background] Flory J, Emanuel E. Interventions to improve research participants' understanding in informed consent for research: a systematic review. JAMA. 2004 Oct 6;292(13):1593-601. doi: 10.1001/jama.292.13.1593. PMID 15467062